CLINICAL TRIAL: NCT01821976
Title: Transtibial Amputation Outcomes Study (TAOS): Comparing Transtibial Amputation With (Ertl) and Without a Tibia-fibula Synostosis Procedure
Brief Title: Transtibial Amputation Outcomes Study
Acronym: TAOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Major Extremity Trauma Research Consortium (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: W8XWH-10-2-0090
Record Dates: First submitted 2013-03-27; First posted 2013-04-01 (Estimated); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Transtibial Amputation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ertl Procedure (Active Comparator): Patients randomized to the Ertl Procedure Arm will receive an amputation very similar to the Burgess Procedure, except the surgeon will perform an additional step to make the cut end of the tibia bone heal to the cut end of the fibula bone with a bone bridge. This bone bridge connects the two bones together.
  Interventions: Procedure: Ertl Procedure
- Burgess Procedure (Active Comparator): Patients randomized to the Burgess Procedure Arm will receive a below the knee amputation where the bone is cut and skin and muscle from the back of the leg are rotated to cover the cut end of your bone. This provides good soft tissue padding to the bone and a good shape to the leg for later fitting of your prosthesis.
  Interventions: Procedure: Burgess Procedure

INTERVENTIONS:
Procedure: Ertl Procedure
  Arms: Ertl Procedure
Procedure: Burgess Procedure
  Arms: Burgess Procedure

SUMMARY:
The goals of the TAOS study is to determine the best procedures for below the knee amputations. There are two different procedures currently used by surgeons around the county: the Erlt procedure and the Burgess procedure. Proponents of the Ertl procedure advocate that the surgical formation of a tibia to fibula bone bridge provides stability, shape and weight bearing capability to the residual limb that result in less pain and better prosthetic fit and alignment. This procedure is popular especially among the military but it's advantages over the Burgess procedure are not well supported by current research. This study aims to compare the two amputation procedures in an adequately powered randomized trial.

DETAILED DESCRIPTION:
High-energy open fractures, blast, gunshot wound and crush injuries to the distal tibia, ankle, hind foot and midfoot are common challenges to military and civilian trauma surgeons (Brown, 2009; Covey, 2002; Ficke, 2007; McGuigan, 2007; Hansen, 2001). Many surgeons believe that an early transtibial amputation provides a better long term functional outcome than limb salvage for these injuries (Hansen, 2001; Myerson, 1994; Sanders, 1992; Turchin,1999; Shawen, 2010;Ellington 2012). If a transtibial amputation is selected as the treatment for the patient, a controversy remains regarding the appropriate amputation technique. Many surgeons advocate for an amputation with a tibia-fibula synostosis technique (Ertl procedure) in young and active patients, believing that this procedure provides a better prosthetic interface, an end bearing capacity and soft tissue stability that improves performance and functional outcomes. (Pinto 2004; Pinzur 2006; Commuri 2010). Others strongly advocate for a standard posterior flap (Burgess procedure) without the synostosis, arguing that patients have similar outcomes with fewer complications and lower costs. (Pinzur 2008; Tindle 2011) To date, the outcomes of the transtibial amputation techniques have not been subjected to an appropriately powered prospective randomized clinical trial.

The primary study objective is to compare functional outcomes and number of revision surgeries to the amputated limb after first amputation for patients undergoing a transtibial amputation and randomized to receive a tibia-fibula synostosis (Ertl procedure) versus a standard posterior flap procedure (Burgess procedure).

The secondary study objectives are to compare levels of impairment for patients undergoing a transtibial amputation and randomized to receive a tibia-fibula synostosis (Ertl procedure) versus a standard posterior flap procedure (Burgess procedure); to compare levels of pain for patients undergoing a transtibial amputation and randomized to receive a tibia-fibula synostosis (Ertl procedure) versus a standard posterior flap procedure (Burgess procedure); and to compare initial hospitalization and overall treatment costs (through the 18 month follow-up) for patients undergoing a transtibial amputation and are randomized to receive a tibia-fibula synostosis (Ertl procedure) versus a standard posterior flap procedure (Burgess procedure). Patients who refuse randomization have the option of participating in a prospective observational study and the type of amputation is decided by the surgeon and patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring a unilateral transtibial amputation following major limb trauma regardless of when the injury occurred
* The injury and its treatment must meet the following criteria:

  * The residual fibula is not fractured or if fractured, is stabilized by internal fixation allowing for either the Ertl or Burgess procedure
  * Proximal tibia/fibula joint is stabilized
  * Soft tissue coverage allows for atypical closure and skin graft <100 cm2
  * Amputation will result in a residual limb that is ≥10 cm from joint line to end of tibia
* Ages 18 and 60 inclusive

Exclusion Criteria:

* At time of consent, patient has a Glasgow Coma Scale (GCS) motor score of 0-4 or a GCS motor score of 5 with a significant traumatic brain injury (defined as an AIS code of 5 or 6)
* Patients with wound closure requiring a free tissue transfer
* Fibula fractures proximal to the tibial bone cut that cannot be stabilized
* Late amputation with presence of one of the following conditions: (i) infection within the zone of injury; (ii) chronic regional pain syndrome; (iii) post-traumatic thrombophlebitis
* Patient has a spinal cord deficit
* Patient has a previous leg or foot amputation or is non-ambulatory pre-injury
* Patient has third degree burns on >10% total surface area affecting the study limb
* Patient has a documented psychiatric disorder
* Patient is unable to speak either English or Spanish
* Severe problems with maintaining follow-up (e.g. patients who are prisoners or homeless at the time of injury or who are intellectually challenged without adequate family support).
* Patient has an amputation to one or both upper extremities (excluding digits)
* Patient is outside hospital's catchment area
* Patient follow-up is planned at another medical center

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 250 (Estimated)
Dates: Start 2013-03; Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Patient Reported Function | 18 Months
  Patient reported function as measured using the Short Form Musculoskeletal Assessment (SMFA) 18 months following amputation
Number of Revision Surgeries | 18 Months
  Number of revision surgeries to the amputated limb within 18 months after the first amputation

SECONDARY OUTCOMES:
Physical Impairment | 18 Months
  Physical impairment will be determined using objective performance measures of agility (4 step square test and Illinois Agility Test), strength and power (sit-to-stand test and timed stair climb), speed (self-selected walking speed and 40 yard shuttle run), postural stability (single leg stance) and overall activity measured using the Step Watch activity monitor
Self Reported Pain | 18 Months
  Pain measured using the Brief Pain Inventory (BPI) questionnaire
Treatment Costs | 18 Months
  Initial hospitalization and overall treatment costs as determined from hospitals bills and data on utilization of outpatient health services

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Reider, MHS, PhD, Study Director — Johns Hopkins University
Locations (23):
- United States (23):
  - University of California San Francisco Medical Center, San Francisco, California
  - University of Miami Ryder Trauma Center, Miami, Florida
  - Florida Orthopaedic Institute- Tampa General Hospital, Tampa, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Eskenazi Health, Indianapolis, Indiana
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - University of Maryland/R Adams Cowley Shock Trauma Medical Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Barnes Jewish Hospital, St Louis, Missouri
  - St. Louis University Medical Center, St Louis, Missouri
  - Carolinas Medical Center, Charlotte, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - MetroHealth Medical Center, Cleveland, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Penn State University M.S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Brown University, Providence, Rhode Island
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - San Antonio Miliary Medical Center, Fort Sam Houston, Texas
  - UT Health: The University of Texas Health Science Center at Houston Medical School, Houston, Texas
  - University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin